CLINICAL TRIAL: NCT05774977
Title: Study on the Use of Broadband Sound to Mitigate Sleep Disruption Due to Aircraft Noise
Brief Title: Broadband Sound and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Civil Aerospace Medical Institute (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 852479
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Noise Exposure
Keywords: Sleep; Cognitive Performance
MeSH Terms: interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: We will investigate participants in 7 groups of 4 subjects each. For six nights following an adaptation night, a different noise condition occurred each night. Each participant of a group was exposed to the same condition in each study night. In this randomization paradigm, each condition will appear in each position exactly once, and will be preceded by each other condition exactly once.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, study personnel and those assessing outcomes will be unaware of order of the exposure conditions. Investigators will only learn about the condition after the start of the sleep period of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pink Noise Only, 50 dBA (BN50) (Experimental): Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on night 1, subjects received the Pink Noise at 50 dBA (BN50) condition once between nights 2 to 7.
  The Pink Noise at 50 dBA (BN50) night consisted of exposure to continuous pink broadband noise throughout the sleep period at a level of 50 A-weighted decibels (dBA).
  For the purposes of blinding, this was Condition A.
  Interventions: Other: Aviation Noise Only (AN); Other: Pink noise only, 50 dBA (BN50); Other: Aviation Noise With Earplugs (AN+EP); Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40); Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50)
- Aviation Noise Plus Pink Noise at 50 dBA (AN+BN50) (Experimental): Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on night 1, subjects received the Aviation Noise + Pink Noise at 50 dBA (AN+BN50) condition once between nights 2-7.
  The Aviation Noise plus Pink Noise, 50 dBA (AN+BN50) night consisted of aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 50 dBA (BN50). The aviation noise (AN) was a pre-programmed recording of 93 sounds including aviation-related noise (e.g. helicopter, sonic boom) and alerting noise (alarm, baby crying), ranging from 45 dB to 65 dB, played during sleep from 2300-0700.
  For the purposes of blinding, this was Condition B.
  Interventions: Other: Aviation Noise Only (AN); Other: Pink noise only, 50 dBA (BN50); Other: Aviation Noise With Earplugs (AN+EP); Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40); Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50)
- Control (CTRL) (Sham Comparator): Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on night 1, subjects received the Control (CTRL) condition once between nights 2 to 7.
  The Control (CTRL) night had no interventions. There was no background broadband noise nor aviation noise, and subjects did not wear earplugs.
  For the purposes of blinding, this was Condition C.
  Interventions: Other: Aviation Noise Only (AN); Other: Pink noise only, 50 dBA (BN50); Other: Aviation Noise With Earplugs (AN+EP); Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40); Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50)
- Aviation Noise Plus Pink Noise at 40 dBA (AN+BN40) (Experimental): Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on night 1, subjects received the Aviation Noise plus Pink Noise at 40 dBA (AN+BN40) condition once between nights 2 to 7.
  The Aviation Noise plus Pink Noise at 40 dBA (AN + BN40) night consisted of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 40 A-weighted decibels (dBA). The aviation noise (AN) was a pre-programmed recording of 93 sounds including aviation-related noise (e.g. helicopter, sonic boom) and alerting noise (alarm, baby crying), ranging from 45 dB to 65 dB, played during sleep from 2300-0700.
  For the purposes of blinding, this was Condition D.
  Interventions: Other: Aviation Noise Only (AN); Other: Pink noise only, 50 dBA (BN50); Other: Aviation Noise With Earplugs (AN+EP); Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40); Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50)
- Aviation Noise (AN) (Experimental): Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on night 1, subjects received the Aviation Noise (AN) condition once between nights 2 to 7.
  The aviation noise (AN) was a pre-programmed recording of 93 sounds including aviation-related noise (e.g. helicopter, sonic boom) and alerting noise (alarm, baby crying), ranging from 45 dB to 65 dB, played during sleep from 2300-0700.
  There was no broadband noise exposure overnight. For the purposes of blinding, this was Condition E.
  Interventions: Other: Aviation Noise Only (AN); Other: Pink noise only, 50 dBA (BN50); Other: Aviation Noise With Earplugs (AN+EP); Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40); Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50)
- Aviation Noise Plus Earplugs (AN+EP) (Experimental): Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on night 1, subjects received the Aviation Noise plus Earplugs (AN+EP) condition once between nights 2 to 7.
  The aviation noise (AN) was a pre-programmed recording of 93 sounds including aviation-related noise (e.g. helicopter, sonic boom) and alerting noise (alarm, baby crying), ranging from 45 dB to 65 dB, played during sleep from 2300-0700. There was no broadband noise exposure.
  For the purposes of blinding, this was Condition F.
  Interventions: Other: Aviation Noise Only (AN); Other: Pink noise only, 50 dBA (BN50); Other: Aviation Noise With Earplugs (AN+EP); Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40); Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50)

INTERVENTIONS:
Other: Aviation Noise Only (AN) — The aviation noise (AN) night will expose subjects to a pre-programmed recording of aviation noise and alerts during sleep from 2300-0700.
Other: Pink noise only, 50 dBA (BN50) — The BN50 night will consist of exposure to continuous pink noise throughout the sleep period at a level of 50 A-weighted decibels (dBA).
Other: Aviation Noise With Earplugs (AN+EP) — The AN + EP night will consist of the aviation noise (AN) exposure with the addition of wearing earplugs overnight.
Other: Aviation Noise With Pink Noise, 40 dBA (AN+BN40) — The AN + BN40 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 40 dBA.
Other: Aviation Noise With Pink Noise, 50 dBA (AN+BN50) — The AN + BN50 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 50 dBA.

SUMMARY:
Sound insulation of bedrooms is expensive and typically only granted to residents living close to the airport. We plan to investigate the effects of various aviation noises on sleep under controlled laboratory conditions and to investigate whether some of the sleep disturbing effects can be mitigated by introducing broadband noise into the bedroom or by wearing earplugs.

DETAILED DESCRIPTION:
The Federal Aviation Administration is interested in investigating inexpensive yet effective methods to mitigate the adverse effects of aviation noise on sleep. The sleep of up to 28 subjects will be monitored with polysomnography and actigraphy over 7 consecutive nights in groups of 4 exposed to various sound conditions (aviation noise; broadband noise; aviation noise plus earplugs; aviation noise plus broadband noise at various decibel [dB] levels). Subjects will fill out surveys, perform cognitive tasks and a hearing test before and after each sleep period. The study will be performed in the Chronobiology Isolation Laboratory (CIL) in the Hospital of the University of Pennsylvania. This newly constructed facility includes 4 acoustically isolated bedrooms and a high-fidelity sound system. Eligible subjects are age 21-50, free of psychiatric conditions that preclude participation, and maintain a self-reported regular sleep schedule of 6-8.5 hours per night as verified by six days of ambulatory actigraphy and daily logs.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects between 21-50 years old
* Free of psychological/psychiatric conditions that preclude participation.
* BMI between 18.5 and 35.
* Self-reported regular sleep schedule; able to maintain their sleep schedule during the course of the study.
* Self-reported sleep duration of 6-8.5 h per night (verified by ambulatory sleep monitoring with wrist actigraphy and daily logs).
* Ability to read/write English.
* Fully vaccinated for or recovered from coronavirus (COVID-19).

Exclusion Criteria:

* Subjects habitually use broadband noise (e.g. white noise machines) to promote sleep at home.
* Hearing loss greater than 25 dB in any frequency band up to 8 kilohertz (kHz).
* History of neurological, psychiatric, or other medical condition that excludes participation.
* Current mania or psychosis.
* Current depression as determined by the Beck Depression Inventory with a score of 17 or greater (Beck, 1996).
* Alcohol or drug abuse in the past year based upon history and urine toxicology screen.
* Excessive alcohol intake (above 21 drinks per week) or binge alcohol consumption (5 or more drinks per day).
* Excessive caffeine consumption (above 650mg/day combining all caffeinated drinks regularly absorbed during the day).
* Current smoker/tobacco user, or using nicotine replacement therapy. Those that have been nicotine-free for 30 days will be included.
* Body Mass Index at or below 18.5 or at or above 35.
* Acute, chronic, or debilitating medical conditions, major Axis I psychiatric illness based on history, physical exam, blood and urine chemistries, and complete blood count (CBC).
* Individuals who self-report a history of recurrent seizures or epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion).
* Cardiovascular, neurological, gastrointestinal, or musculoskeletal problems that exclude participation.
* Major controlled or uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure, cancer, chronic obstructive pulmonary disease (COPD), respiratory failure or insufficiency, cardiac arrhythmia, or patients requiring oxygen therapy (as determined by self-report).
* Currently working night, swing, split or rotating shift.
* Current use or use of within the past month of a prescription or over-the-counter sleep medication or stimulant; use of psychoactive medication (based on self-report and review with a study clinician).
* Pregnant or currently breast feeding.
* Prior history or diagnosis of any sleep disorder including Obstructive Sleep Apnea (OSA) (AHI at or above 15 events/hour) from ambulatory or in lab polysomnography; Restless legs syndrome or periodic limb movement disorder; Insomnia; Parasomnia; High Risk of OSA based on Stop-Bang Questionnaire (yes on at least 4 of 8 questions); High Risk of Restless Legs Syndrome (RLS) based on Cambridge-Hopkins Screening questionnaire; High Risk of Insomnia based on Insomnia Severity Index (score of 22 or higher).
* Individuals who self-report severe contact dermatitis or allergy to silicone, nickel or silver.
* Planned travel across more than one time zone one month prior to and/or during the anticipated period of the study.
* Intentional naps during the week.
* Positive COVID-19 test at prescreening.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Basner, MD, PhD, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Public project data files will be available via the National Transportation Library (NTL). Personally Identifiable Information (PII) will not be publicly available. Sensitive data that cannot be de-identified will be posted to secure government databases, such as posting of genetic sequence data in NIH's database of Genotypes and Phenotypes (dbGAP) (www.ncbi.nlm.nih.gov/gap/), where appropriate and in accordance with institutional review board (IRB) guidance and federal regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data files will be available one year after the project end date.
Access Criteria: People requesting the data will have to fulfill the access criteria set by the respective database.

REFERENCES:
- [Background] Huang HW, Zheng BL, Jiang L, Lin ZT, Zhang GB, Shen L, Xi XM. Effect of oral melatonin and wearing earplugs and eye masks on nocturnal sleep in healthy subjects in a simulated intensive care unit environment: which might be a more promising strategy for ICU sleep deprivation? Crit Care. 2015 Mar 19;19(1):124. doi: 10.1186/s13054-015-0842-8. PMID 25887528
- [Background] Riedy SM, Smith MG, Rocha S, Basner M. Noise as a sleep aid: A systematic review. Sleep Med Rev. 2021 Feb;55:101385. doi: 10.1016/j.smrv.2020.101385. Epub 2020 Sep 9. PMID 33007706
- [Background] Watson NF, Badr MS, Belenky G, Bliwise DL, Buxton OM, Buysse D, Dinges DF, Gangwisch J, Grandner MA, Kushida C, Malhotra RK, Martin JL, Patel SR, Quan SF, Tasali E. Recommended Amount of Sleep for a Healthy Adult: A Joint Consensus Statement of the American Academy of Sleep Medicine and Sleep Research Society. Sleep. 2015 Jun 1;38(6):843-4. doi: 10.5665/sleep.4716. PMID 26039963
- [Background] Basner M, McGuire S. WHO Environmental Noise Guidelines for the European Region: A Systematic Review on Environmental Noise and Effects on Sleep. Int J Environ Res Public Health. 2018 Mar 14;15(3):519. doi: 10.3390/ijerph15030519. PMID 29538344
- [Background] Basner M, Babisch W, Davis A, Brink M, Clark C, Janssen S, Stansfeld S. Auditory and non-auditory effects of noise on health. Lancet. 2014 Apr 12;383(9925):1325-1332. doi: 10.1016/S0140-6736(13)61613-X. Epub 2013 Oct 30. PMID 24183105
- [Derived] Basner M, Smith MG, Cordoza M, Kayser MS, Carlin M, Ecker AJ, Gilad Y, Park-Chavar S, Rennie K, Schneller V, Walsh S, Shou H, Cao Q, Younes M, Aeschbach D, Jones CW. Efficacy of pink noise and earplugs for mitigating the effects of intermittent environmental noise exposure on sleep. Sleep. 2026 Feb 2:zsag001. doi: 10.1093/sleep/zsag001. Online ahead of print. PMID 41627391

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was designed to expose all subjects to the six noise conditions after an adaptation night. However, the order in which subjects experienced each condition varied, resulting in seven different condition sequences. Subjects were assigned to a study group with up to 4 total participants, where each participant experienced the same condition sequence. A total of 27 subjects were enrolled and assigned to one of the seven sequences.
Groups:
- Noise Condition: This study uses within-subject comparison. For each subject, the order of noise conditions for each of the six nights following an adaptation night will be randomized. All subjects will receive all noise conditions.
  Please refer to the study design and protocol for additional information.
  A. Pink noise, 50 dBA only (BN50): The BN50 night consisted of exposure to continuous pink noise throughout the sleep period at a level of 50 A-weighted decibels (dBA).
  B. Aviation noise plus pink noise 50 dBA (AN+BN50): The AN + BN50 night consisted of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 50 dBA.
  C. Control night (CTRL) without noise exposure and without earplugs.
  D. Aviation noise plus pink noise 40 dBA (AN+BN40): The AN + BN40 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 40 dBA.
  E. Aviation Noise Only (AN): The aviation noise (AN) exposure was a pre-programmed recording of 93 sounds, including aviation-related noises (e.g. helicopter, sonic boom) and alerting noise (alarm, baby crying) with a range between 45 dB to 65 dB, played during sleep from 2300-0700.
  F. Aviation noise plus earplugs (AN+EP): The AN + EP night consist of the aviation noise (AN) exposure with the addition of wearing earplugs during the sleep period.
Period: Overall Study
Arm/Group | Noise Condition
Started | 27
Pink Noise, 50 dBA (BN50) | 25
Aviation Noise Plus Pink Noise 50 dBA (AN+BN50) | 24 (One subject withdrew after night 5. Their data was included in analysis of the conditions they were exposed to. As this condition occurred after their withdrawal, they were not included in the AN+BN50 analysis.)
Control Night (CTRL) | 21 (In Group 3, the PSG system failed in three out of four subjects on night 2, which was planned to be the Control condition. It was thus decided by the PI to repeat the Control condition on a following night (night 6), which resulted in Group 3 not receiving the Aircraft noise + ear plugs (condition F) exposure.)
Aviation Noise Plus Pink Noise 40 dBA (AN+BN40) | 24 (One subject withdrew after night 5. Their data was included in analysis of the conditions they were exposed to. As this condition occurred after their withdrawal, they were not included in the AN+BN40 analysis.)
Aviation Noise Only (AN) | 25
Aviation Noise Plus Earplugs (AN+EP) | 25
Completed | 25
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: While 27 subjects were enrolled in the study, 25 were used for final analysis. Two subjects (N=2) were excluded from analysis due to withdrawing from the study: 1 subject withdrew from Group 2 after night 2, and 1 subject withdrew from Group 7 after night 3. An additional subject withdrew after experiencing 4 of the 6 noise conditions, and therefore their data were included in analysis of the noise conditions to which they were exposed.
Groups:
- Group 1: A B C D E F: Subjects in Group 1 experienced the conditions in this order: A B C D E F.
- Group 2: B D A F C E: Subjects in Group 2 experienced the conditions in this order: B D A F C E.
- Group 3: C A E B C D: Subjects in Group 3 were scheduled to experience the conditions in this order: C A E B F D. However, the PSG system failed in three out of four subjects in study night 2. Therefore, it was decided by the PI to rerun the night 2 exposure (condition C) on night 6. In doing so, the condition originally planned for night 6 (condition F) was removed from this study sequence, and Group 3 subjects did not experience the condition F exposure.
- Group 4: D F B E A C: Subjects in Group 4 experienced the conditions in this order: D F B E A C.
- Group 5: E C F B D A: Subjects in Group 5 were scheduled to experience the conditions in this order: E C F A D B. However, due to an inadvertent selection of the audio sequence on night 5, the file for night 7 was played on night 5. Therefore, the noise conditions originally planned for night 5 and 7 were switched in order to expose subjects to all noise conditions.
- Group 6: F E D C B A: Subjects in Group 6 experienced the conditions in this order: F E D C B A.
- Group 7: C D E A F B: Subjects in Group 7 experienced the conditions in this order: C D E A F B.
- Total: Total of all reporting groups
Arm/Group | Group 1: A B C D E F | Group 2: B D A F C E | Group 3: C A E B C D | Group 4: D F B E A C | Group 5: E C F B D A | Group 6: F E D C B A | Group 7: C D E A F B | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject withdrew from Group 2 and was excluded from analysis. One subject withdrew from Group 7 and was excluded from analysis.
  years
    number analyzed (Participants) | 4 | 3 | 4 | 3 | 4 | 4 | 3 | 25
    (all) | 24.25 (1.71) | 30 (9.85) | 30 (2.94) | 26 (4.36) | 28.75 (6.55) | 28.5 (7.85) | 33 (6.56) | 28.54 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 2 | 2 | 2 | 3 | 19
  Male | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
  White | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 7
  More than one race | 2 | 2 | 2 | 0 | 2 | 0 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Slow Wave Sleep and Rapid Eye Movement (N3 + REM)
Description: Combined time spent in sleep stages N3 and REM in minutes, as measured by polysomnography (PSG).
Time Frame: Days 2-7
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Groups:
- Aviation Noise Only: Aviation Noise Only (AN): The aviation noise (AN) night will expose subjects to a pre-programmed recording of aviation noise during sleep from 2300-0700.
- Pink Noise Only (50 dBA): Pink noise, 50 dBA only (BN50): The BN50 night will consist of exposure to continuous pink noise throughout the sleep period at a level of 50 A-weighted decibels (dBA).
- Aviation Noise With Earplugs: Aviation noise plus earplugs (AN+EP): The AN + EP night will consist of the aviation noise (AN) exposure with the addition of wearing earplugs overnight.
- Aviation Noise With Pink Noise, 40 dBA: Aviation noise plus white noise 40 dBA (AN+BN40): The AN + BN40 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 40 dBA.
- Aviation Noise With Pink Noise, 50 dBA: Aviation noise plus white noise 50 dBA (AN+BN50): The AN + BN50 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 50 dBA.
- Control: Control Night (CTRL): Control night (CTRL) without noise exposure and without earplugs.
Arm/Group | Aviation Noise Only | Pink Noise Only (50 dBA) | Aviation Noise With Earplugs | Aviation Noise With Pink Noise, 40 dBA | Aviation Noise With Pink Noise, 50 dBA | Control
Number analyzed (Participants) | 25 | 25 | 21 | 24 | 24 | 25
Minutes | 188.5532184 [172.8271298 to 204.279307] | 195.9798771 [180.1286092 to 211.831145] | 209.51862074703 [193.2405983 to 225.7966432] | 176.4599674 [160.6090035 to 192.3109313] | 174.2895997 [158.4417133 to 190.1374861] | 219.0943443 [203.4591503 to 234.7295384]

2. Secondary Outcome: Cognition Efficiency
Description: Efficiency scores from 10 brief cognitive tasks are generated from accuracy & speed of reaction/responding, represented here by standardized effect sizes, where higher scores indicate better performance. Test scores were adjusted for practice and stimulus set effects, and z-transformed based on average and standard deviation across all tests taken. Accuracy and speed across cognitive domains were calculated by averaging z-scores across the 10 tests, then averaged to calculate an efficiency metric.
  Scores between -0.2 and +0.2 suggest no effect on efficiency (0=population mean).
  Between -0.2 and -0.5 suggests a small negative effect (i.e. slightly less efficient).
  Between -0.5 and -0.8 suggests a moderate negative effect. Scores below -0.8 suggest a large negative effect. Between 0.2 and 0.5 suggests a small positive effect. Between 0.5 and 0.8 suggests a moderate positive effect. Scores above 0.8 suggest a large positive effect (i.e. significantly more efficient).
Time Frame: Days 2-7
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Aviation Noise Only | Pink Noise Only (50 dBA) | Aviation Noise With Earplugs | Aviation Noise With Pink Noise, 40 dBA | Aviation Noise With Pink Noise, 50 dBA | Control
Number analyzed (Participants) | 25 | 25 | 21 | 24 | 24 | 25
Z-score | -0.064223254075 (0.065476995) | -0.080820342 (0.065961006) | -0.002037537 (0.067457746) | -0.005021343 (0.065934126) | -0.02031753 (0.065473068) | -0.061364516 (0.064361916)

3. Secondary Outcome: Cognition Speed
Description: A single variable representing response time across 10 Cognitive tasks that cover a range of cognitive domains with known cerebral representation. Test scores were adjusted for practice and stimulus set effects, and z-transformed based on average and standard deviation across all tests taken. Speed across cognitive domains was calculated by averaging z-scores across the 10 tests. Higher scores reflect faster speed.
  Scores between -0.2 and +0.2 suggest no effect on speed (0=population mean). Between -0.2 and -0.5 suggests a small negative effect (i.e. slightly slower). Between -0.5 and -0.8 suggests a moderate negative effect. Scores below -0.8 suggest a large negative effect (i.e. significantly slower). Between 0.2 and 0.5 suggests a small positive effect (i.e. slightly faster). Between 0.5 and 0.8 suggests a moderate positive effect. Scores above 0.8 suggest a large positive effect (i.e. significantly faster).
Time Frame: Days 2-7
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Aviation Noise Only | Pink Noise Only (50 dBA) | Aviation Noise With Earplugs | Aviation Noise With Pink Noise, 40 dBA | Aviation Noise With Pink Noise, 50 dBA | Control
Number analyzed (Participants) | 25 | 25 | 21 | 24 | 24 | 25
z-score | -0.133247423 (0.115983876) | -0.144315479 (0.116338083) | -0.057069789 (0.117437672) | -0.056543403 (0.116319131) | -0.078872577 (0.115981035) | -0.08897121 (0.115186663)

4. Secondary Outcome: Cognition Accuracy
Description: A single variable representing response time across 10 Cognitive tasks that cover a range of cognitive domains with known cerebral representation. Test scores were adjusted for practice and stimulus set effects, and z-transformed based on average and standard deviation across all tests taken. Accuracy across cognitive domains was calculated by averaging z-scores across the 10 tests. Higher scores reflect better accuracy.
  Scores between -0.2 and +0.2 suggest no effect on accuracy (0=population mean). Between -0.2 and -0.5 suggests a small negative effect (i.e. slightly less accurate).
  Between -0.5 and -0.8 suggests a moderate negative effect. Scores below -0.8 suggest a large negative effect (i.e. significantly less accurate).
  Between 0.2 and 0.5 suggests a small positive effect (i.e. slightly more accurate).
  Between 0.5 and 0.8 suggests a moderate positive effect. Scores above 0.8 suggest a large positive effect (i.e. significantly more accurate).
Time Frame: Days 2-7
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Aviation Noise Only | Pink Noise Only (50 dBA) | Aviation Noise With Earplugs | Aviation Noise With Pink Noise, 40 dBA | Aviation Noise With Pink Noise, 50 dBA | Control
Number analyzed (Participants) | 25 | 25 | 21 | 24 | 24 | 25
z-score | 0.004818355 (0.082094556) | -0.016730648 (0.082952084) | 0.055614609 (0.085599407) | 0.04713328 (0.082902765) | 0.038223035 (0.082087524) | -0.035636712 (0.080077528)

5. Secondary Outcome: Driving Simulator Standard Deviation of Lane Position
Description: The standard deviation of lane position reflects the extent (in feet) to which participants "swerve" within the lane in a virtual driving simulator, often used to investigate the effects of impairment on driving performance, where higher values represent worse performance.
Time Frame: Days 2-7
Measure: Least Squares Mean (Standard Deviation); unit: feet
Arm/Group | Aviation Noise Only | Pink Noise Only (50 dBA) | Aviation Noise With Earplugs | Aviation Noise With Pink Noise, 40 dBA | Aviation Noise With Pink Noise, 50 dBA | Control
Number analyzed (Participants) | 25 | 25 | 21 | 24 | 24 | 25
feet | 1.40658463 (0.088697515) | 1.394516627 (0.08888539) | 1.340740078 (0.089469215) | 1.425292912 (0.088875405) | 1.359432551 (0.088696012) | 1.377041493 (0.08827651)

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events over the course of their in-laboratory participation, starting with the adaptation night through the completion of the six overnight conditions, for a period of 7 nights.
Groups:
- Group 1: A B C D E F; Group 2: B D A F C E; Group 3: C A E B C D; Group 4: D F B E A C; Group 5: E C F B D A; Group 6: F E D C B A; Group 7: C D E A F B: Subjects were exposed to six different conditions during a sleep opportunity period from 2300-0700. After an adaptation night with no interventions on Night 1, subjects received the exposure sequence listed under Arm/Group Title.
  A = Pink noise, 50 dBA only (BN50): The BN50 night will consist of exposure to continuous pink noise throughout the sleep period at a level of 50 A-weighted decibels (dBA).
  B = Aviation noise plus white noise 50 dBA (AN+BN50): The AN + BN50 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 50 dBA.
  C = Control Night (CTRL): Control night (CTRL) without noise exposure and without earplugs.
  D = Aviation noise plus white noise 40 dBA (AN+BN40): The AN + BN40 night will consist of the aviation noise (AN) exposure with the addition of continuous pink noise throughout the sleep period at a level of 40 dBA.
  E = Aviation Noise Only (AN): The aviation noise (AN) night will expose subjects to a pre-programmed recording of aviation noise during sleep from 2300-0700.
  F = Aviation noise plus earplugs (AN+EP): The AN + EP night will consist of the aviation noise (AN) exposure with the addition of wearing earplugs overnight.
Arm/Group | Group 1: A B C D E F | Group 2: B D A F C E | Group 3: C A E B C D | Group 4: D F B E A C | Group 5: E C F B D A | Group 6: F E D C B A | Group 7: C D E A F B
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/77/NCT05774977/Prot_SAP_002.pdf
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT05774977/ICF_001.pdf